CLINICAL TRIAL: NCT00299793
Title: Observational Study of Lamotrigine
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: 01.08.110
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Epilepsy
Keywords: Epilepsy; Quality of life
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess efficacy, safety and tolerability of lamotrigine as used in a natural clinical setting, to examine the positive effects of lamotrigine, and the reasons why some patients choose to continue or discontinue lamotrigine.

DETAILED DESCRIPTION:
There have been numerous randomized, double-blind controlled trials demonstrating the value of lamotrigine in the treatment of seizures. However, randomized trials take place in artificial experimental conditions with many restrictions imposed. There hasn't been much focus on positive effects on the patient, such as improvement in mood and level of alertness related to the drug. Other factors related to quality of life that affect the decision to continue or discontinue the drug are also important. Anecdotal experience suggests that lamotrigine is associated with increased alertness, enhanced energy levels and improved general sense of well-being. Observational studies that promote awareness of such distinguishing features and other aspects of efficacy are essential for guiding decision-making when prescribing anti-epileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are about to be prescribed lamotrigine as an appropriate treatment for their epileptic disorder

Exclusion Criteria:

* Patients with mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ettinger, MD, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States